CLINICAL TRIAL: NCT03588455
Title: Pronostic Impact of Flow Fraction Reserve on Intermediate Stenoses
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: FFR
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Coronary Stenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The intermediate coronary stenoses defined by a degree of stenosis from 40 to 70 % are frequent. The Flow Fraction Reserve (FFR), realized during coronarography, is an hemodynamic evaluation by the functional impact measuring the loss of load in upstream / approval of the stenosis inthe basal state and in situation of hyperemia led by adenosine. Further to the study FAME, the threshold of definition of the significant character of one Stenosis was fixed for a value of FFR = 0,80. However, the impact forecasts intermediate values badly known rest.

We hypothetized that coronary stenosis associated with borderline values of FFR 0.81-0.85 were associated with a higher rate of clinical events than those with a FFR >0.85

ELIGIBILITY:
Inclusion Criteria:

* patient with FFR> 0,80 between september 2012 till december 2016

Exclusion Criteria:

* refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient underwent FFR during angiography between 2012 september and december 2016
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Composite outcome | 3 years
  cardiovascular mortality or acute coronary syndrom or revascularization or cardiovascular rehospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: AZZAZ P Sofien, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided